CLINICAL TRIAL: NCT00005950
Title: Phase II Study of 506U78 (NSC #686673) for Patients With Relapsed or Refractory Indolent B-Cell or Peripheral T-Cell Lymphoma
Brief Title: 506U78 in Treating Patients With Recurrent or Refractory Non-Hodgkin's Lymphoma or T-cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02339; ID99-208; N01CM17003 (NIH); CDR0000067894 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-07-05; First posted 2004-04-20 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Angioimmunoblastic T-cell Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Nodal Marginal Zone B-cell Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Splenic Marginal Zone Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Immunoblastic Lymphadenopathy; Lymphoma, B-Cell, Marginal Zone; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — nelarabine

ARMS (1):
- Treatment (Experimental): Patients receive 506U78 IV over 2 hours on days 1, 3, and 5. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: nelarabine

INTERVENTIONS:
Drug: nelarabine — Given IV
  Other Names: 506U78; Arranon; GW506U78

SUMMARY:
Phase II trial to study the effectiveness of 506U78 in treating patients who have recurrent or refractory non-Hodgkin's lymphoma or T-cell lymphoma. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the response rate, failure-free survival, and progression-free survival of patients with recurrent or refractory indolent B-cell non-Hodgkin's lymphoma or peripheral T-cell lymphoma when treated with 506U78.

II. Assess the pharmacokinetics and toxicity of this treatment in these patients.

OUTLINE:

Patients receive 506U78 IV over 2 hours on days 1, 3, and 5. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed or refractory indolent B-cell non-Hodgkin's lymphoma or peripheral T-cell lymphoma

  * Indolent B-cell lymphoma will include Waldenström's macroglobulinemia, lymphoplasmacytoid lymphoma small lymphocytic lymphoma, marginal zone lymphoma, and follicular small cleaved-cell or mixed cell lymphoma; patients with prior or concurrent evidence of transformation to large cell lymphoma or with follicular large cell lymphoma are ineligible
  * Peripheral T-cell lymphoma will include all entities described in the REAL classification; patients with B-cell ALCL are ineligible; patients with cutaneous T-cell lymphoma and all its variants and/or histologic transformation of cutaneous T-cell lymphoma are not eligible for this protocol, because they will be instead eligible for a separate protocol
  * Relapsed peripheral T-cell lymphomas include all those achieving and maintaining a complete or partial response during initial therapy; refractory includes those achieving all other responses during initial therapy; since the response rate of indolent B-cell lymphomas to up-front therapy exceeds 90% this distinction is not meaningful there
* No more than 2 prior chemotherapy and one prior immunotherapy regimens; if chemoimmunotherapy was used, the limit will be 3 prior regimens
* Performance status =< 2 Zubrod
* Staging work-up within 3 weeks and bidimensionally measurable disease
* No anti-cancer treatment within the past three weeks
* ANC >= 1,000/ul; may be included if in the judgment of the study chairman lower counts are explained by marrow or splenic involvement by lymphoma
* Platelets >= 100,000/ul; may be included if in the judgment of the study chairman lower counts are explained by marrow or splenic involvement by lymphoma
* Bilirubin =< 1.5 x normal
* SGPT =< 2.5 x normal values
* Estimated endogenous creatinine clearance > 50 ml/min
* HIV negative; the patients are excluded because the expected opportunistic infections will render study toxicity difficult to interpret; in addition the possible effects of 506U78 on CD4 cells may be dangerous to these patients; furthermore, indolent B-cell lymphomas and aggressive peripheral T-cell lymphomas are extremely rare in the setting of HIV infection
* No active CNS disease
* No other malignancy within the last 5 years, except basal cell carcinoma of the skin or in-situ cervical carcinoma treated with curative intent
* Females must not be pregnant or breast feeding and must be practicing adequate contraception; this is because 506U78 may be harmful to the developing fetus and nursing newborn or infant
* No preexisting sensory or motor neuropathy of grade ≥ 2, no history of seizures
* No prior stem cell or bone marrow transplantation; no prior 506U78
* All patients, including women or members of a minority that fulfill criteria for study entry will be eligible for treatment; no one fulfilling all these criteria for entry will be denied treatment solely on the basis of sex or minority status
* Patients with medical, psychiatric, or social conditions that make compliance with treatment or follow-up unlikely are not eligible
* No history of symptomatic cardiac dysfunction or pericardial effusion

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2000-04; Primary Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Response rate (RR), defined as CR + PR | Up to 5 years

SECONDARY OUTCOMES:
Failure-free survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Andre Goy, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States